CLINICAL TRIAL: NCT02460705
Title: Fecal Microbiota Transplant for Inflammatory Bowel Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Najwa Elnachef, Assistant Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-16617
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IBD patients receiving FMT (Experimental): IBD patients receiving biologically active human fecal material sourced from OpenBiome. The physician will administer 250 mL of the fecal suspension in aliquots of 50-60 mL, through the endoscope. The material will be delivered to the most proximal point of insertion.
  Interventions: Drug: Biologically active human fecal material, OpenBiome

INTERVENTIONS:
Drug: Biologically active human fecal material, OpenBiome — Fecal microbiota transplant

SUMMARY:
Currently enrolling only patients with Ulcerative Colitis. Enrollment and experimental treatment of patients with Crohn's Disease stopped for a safety evaluation.

This is a prospective, open label pilot study in which patients with symptoms of Inflammatory bowel disease will receive FMT therapy delivered via colonoscopy.

The investigators hypothesize that FMT is a safe and effective treatment for patients with inflammatory bowel disease. The aims are:

1. To determine if symptoms of inflammatory bowel disease can be successfully treated by Fecal Microbial Transplantation.
2. To determine if endoscopic appearance of colon or ileum improves following treatment by Fecal Microbial Transplantation.

DETAILED DESCRIPTION:
Currently enrolling only patients with Ulcerative Colitis. Enrollment and experimental treatment of patients with Crohn's Disease stopped for a safety evaluation.

This is a prospective, open label pilot study in which patients with symptoms of acute or chronic inflammatory bowel disease will receive FMT therapy delivered via colonoscopy.

Number of Subjects:

This study will aim to enroll approximately 60 patients with inflammatory bowel disease.

All patients who have IBD will be evaluated at the UCSF Center for Inflammatory Bowel Disease. Patients who are eligible for the study will be identified during these regularly scheduled clinic visits. Patients who express interest will be set up for a meeting with a clinical research coordinator who will go over the study in detail and will obtain informed consent.

Prior to the FMT procedure stool samples will be checked for ova and parasites, C. difficile toxin and fecal calprotectin. Serum tests will include erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), Anti-nuclear antibodies (ANA), complete blood cell count, HIV, screening for Hepatitis A, B, C (hep A IgM, hep B surface antigen and antibody, Hep C antibody), and creatinine. 8 days before treatment, patients will take a 5 day course of rifaximin that is discontinued 3 days before FMT treatment.

Patients with IBD will undergo colonoscopy, which is considered part of standard of care for patients with ongoing inflammation and is not considered a study procedure. The colonoscopies will be done in the endoscopic units at Mt. Zion, Parnassus and/or Mission Bay. During this procedure the fecal transplant will take place. For FMT, 250 cc of FMT material (previously screened stool from OpenBiome) will be administered via the endoscope. The scope will then be withdrawn and the patient will recover in the endoscopy unit as per protocol.

Patients who have undergone FMT for IBD will be called the next day to ensure no adverse events have occurred. Patients will be scheduled for a second FMT treatment and a follow up clinic visit 4 weeks after the inital FMT procedure. Patients will be contacted by phone 24 hours, 1 week, 1 month and and then every 3 months for 3 years after FMT treatment. A 6 month colonoscopy will be done to check for mucosal healing.

During each FMT procedure and the 6 month colonoscopy up to a total of 6 ileum and rectosigmoid biopsies will be obtained. In addition the investigators will collect research blood samples before the initial procedure, 1 and 6 months after the initial FMT treatment.

One week after the second FMT treatment, patients will be given the option to enroll in a 6 week, once per week FMT capsule therapy to be administered at a 1 hour clinic visit. Patients who receive capsules will be called the following to to ensure no adverse events have occurred.

Study participants will be asked to submit a stool sample prior to treatment, one month after treatment and then after that every 3 months after treatment up to 1 year in duration for a total of 6 samples. Study participants will also be administered a patient survey to assess their clinical outcomes/symptoms prior to treatment and again 1 month after receiving treatment. In addition, all patients will receive a phone call 24 hours, 1 week, 1 month and and then every 3 months for 3 years after FMT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of Ulcerative Colitis confirmed by endoscopy and pathology and with a Mayo clinic ulcerative colitits disease activity score of 6 or greater.
* Concurrent therapies with mesalamine, immunomodulators, corticosteroids and biologic agents will be allowed to continue during study.

Exclusion Criteria:

* Female patients who are pregnant.
* Patients with severe immunosuppression (absolute neutrophil count < 1000 or CD4 count <200).
* Patients with untreated enteric infection.
* Patients with colon cancer or dysplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12-20 (Actual); Study Completion 2017-11-04 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of IBD | 4 weeks
  In order to assess clinical improvement of IBD, patients will be scheduled for a 4 week post-FMT treatment clinic visit to assess patient symptoms.

SECONDARY OUTCOMES:
Efficacy of FMT treatment | 4 weeks
  Patients will complete a survey both before and 4 weeks after treatment to evaluate the efficacy of FMT treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Division of Gastroenterology at Mount Zion, San Francisco, California, United States

REFERENCES:
- [Derived] Gutin L, Piceno Y, Fadrosh D, Lynch K, Zydek M, Kassam Z, LaMere B, Terdiman J, Ma A, Somsouk M, Lynch S, El-Nachef N. Fecal microbiota transplant for Crohn disease: A study evaluating safety, efficacy, and microbiome profile. United European Gastroenterol J. 2019 Jul;7(6):807-814. doi: 10.1177/2050640619845986. Epub 2019 Apr 20. PMID 31316785